CLINICAL TRIAL: NCT04400357
Title: Robotic Versus Open Pancreaticoduodenectomy for Pancreatic and Periampullary Tumors: A Multicenter Phase III Non-Inferiority Randomized Controlled Trial
Brief Title: Robotic Versus Open Pancreaticoduodenectomy for Pancreatic and Periampullary Tumors
Acronym: PORTAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Intuitive Surgical (Industry)
Responsible Party: Principal Investigator, JIABIN JIN, Attending Surgeon, Pancreatic Disease Center, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2020-93
Record Dates: First submitted 2020-05-10; First posted 2020-05-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Adenocarcinoma; Pancreatic Cysts; Pancreatic Endocrine Tumors; Chronic Pancreatitis; Cholangiocarcinoma, Extrahepatic; Ampullary Adenocarcinoma; Duodenal Adenocarcinoma
Keywords: pancreaticoduodenectomy; Whipple; robotic; daVinci; pancreatic cancer; outcomes; pancreatectomy; functional recovery; complications; recurrence; circulating tumor DNA; perioperative inflammation
MeSH Terms: conditions — Pancreatic Cyst; Pancreatitis, Chronic; Cholangiocarcinoma; Pancreatic Neoplasms; Recurrence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Robotic pancreaticoduodenectomy (Experimental): Patients randomized in this arm will undergo a robotic pancreaticoduodenectomy.
  Interventions: Procedure: Robotic pancreaticoduodenectomy
- Open pancreaticoduodenectomy (Active Comparator): Patients randomized in this arm will undergo a routine open pancreaticoduodenectomy.
  Interventions: Procedure: Open pancreaticoduodenectomy

INTERVENTIONS:
Procedure: Robotic pancreaticoduodenectomy — Patients in this arm will undergo a pancreaticoduodenectomy with robotic-assisted techonology.
  Arms: Robotic pancreaticoduodenectomy
Procedure: Open pancreaticoduodenectomy — Patients in this arm will undergo an open pancreaticoduodenectomy which is the standard surgical approach.
  Arms: Open pancreaticoduodenectomy

SUMMARY:
This multicenter randomized trial aims to primarily assess and compare the functional recovery of patients who undergo open versus robotic pancreaticoduodenectomy for benign and malignant lesions of the head of the pancreas.

DETAILED DESCRIPTION:
The PORTAL trial is a Phase 3 multicenter non-inferiority randomized controlled trial that aims to address the question of feasibility and efficacy of the robotic minimally invasive approach in pancreaticoduodenectomy.

In the past 10 years there has been an increasing number of retrospective series from major centers for pancreatic surgery worldwide, that demonstrate similar and occasionally improved postoperative outcomes in patients who undergo a robotic pancreaticoduodenectomy (Whipple). The benefits of this minimally invasive approach appear to be decreased intraoperative estimated blood loss, lower postoperative pain levels and smaller length of hospital stay, whereas postoperative complications rates are comparable with the standard open approach.

This trial is conducted in multiple major centers for pancreatic surgery (open and robotic) in China and aims to address these questions in a prospective fashion. All eligible patients who present to these centers within the study period will be randomized in a 1:1 ratio to either of the two arms (open vs. robotic). Patients enrolled in the study will be blinded regarding the type of the procedure by application of identical wound dressings at the trocar sites and the open incision. Patients will be followed up closely and will be evaluated routinely for quality of life parameters for a period of at least 2 years postoperatively. Additionally, patients who undergo surgery in either arm for pancreatic adenocarcinoma will also be evaluated for time to adjuvant chemotherapy postoperatively, as well as recurrence and survival data.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication for elective pancreaticoduodenectomy for malignant, premalignant, and symptomatic benign disease in the pancreatic and periampullary region
* Performance status of 0/1 (assessed based on comorbidities using the Karnofsky score and Malnutrition Universal Screening Tool score among others, especially for patients with malignant disease)
* Imaging with computed tomography and/or MRI pancreas performed within 8 weeks for benign and 4 weeks for malignant disease; for the latter tumor staging with MRI liver, CT chest, and Cancer Antigen 19-9 is also mandatory.

Exclusion Criteria:

* Body mass index > 35 kg/m2
* Pregnancy
* Previous history of major abdominal surgery
* Requirement for multivisceral resection (additional surgical resection)
* Preoperative chemotherapy and/or radiotherapy (for patients with pancreatic adenocarcinoma)
* Involvement of major regional vessels by the tumor (portal and superior mesenteric vein, superior mesenteric artery, hepatic artery, celiac artery) as defined by the borderline resectable and locally advanced nomenclature

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Time to functional recovery postoperatively | From date of surgery to date of functional recovery as described, assessed up to 90 days.
  Daily evaluation of patient postoperative course will take place by the nursing and medical staff and will be documented by the study coordinators. Postoperative criteria that need to be fulfilled independently to achieve functional recovery status are the following:
  * Discontinuation of intravenous or subcutaneous analgesia and preservation of adequate control levels (pain score)
  * Early ambulation and restoration of mobility to an independent level (or to preoperative level if previously impaired)
  * Ability to maintain sufficient oral caloric intake as defined by institutional dietitian services, without intravenous fluid support
  * No clinical signs of active abdominal infection affecting the patient's performance status: absence of fever, white cell count and C-reactive protein decreasing towards normalization. The patient can be in oral antibiotics.

SECONDARY OUTCOMES:
Intraoperative blood loss | During surgery
  Comparison of estimated blood loss (in ml)
Operative time | During surgery
  Comparison of operative time (in minutes, from first incision to skin closure)
Percentage of patients with pancreatic adenocarcinoma who achieve administration of adjuvant chemotherapy at 8 weeks postoperatively | Postoperative Day 1 to Day 56
  The number of patients who are fit and well to initiate adjuvant chemotherapy at the 8-week mark after the operation will be documented and compared between the two arms
Postoperative complication rates and associated interventions | Postoperative Day 1 to Day 30
  Comparison of post-pancreatectomy morbidity between the two surgical approaches, that focus on:
  * Pancreatic fistula
  * Bile leak
  * Chyle leak
  * Delayed gastric emptying
  * Surgical site infection
  * Postoperative pancreatitis
  * Postoperative hemorrhage
  * Surgical site infections
  * Other complications Additional documentation of re-intervention (radiological, endoscopic, or surgical) and re-admission rates, as well as postoperative hospital and ICU length of stay (time to discharge)
Postoperative mortality | Postoperative Day 1 to Day 90
  Comparison of mortality rates as a result of the pancreaticoduodenectomy in each arm
Quality of life measurements | Postoperative Day 1 to Day 90
  For assessment of postoperative quality of life (QoL) improvement, patients will be evaluated with the established EuqoQol EQ-5D-5L questionnaire, which is a self-reported assay focusing on five parameters: Pain/discomfort, anxiety/depression, usual activities, self-care, and mobility. Each of the five aforementioned parameters is scored from 0 to 5 (no issue, slight problem, moderate problem, severe problem, unable); patients also score independently their health status on a scale numbered from 0 to 100; 100 means the best health they can imagine, and 0 the worst.
  Answered questionnaires will be collected on postoperative days 1, 3, 5, 7, and afterwards every week until day 30. QoL evaluation will terminate at Day 90.
Margin resection status (R) in patients with pancreatic adenocarcinoma | During surgery
  In a sub-cohort of patients with pancreatic adenocarcinoma, the margin resection status (R) will be assessed and compared: R0 is defined as presence of tumor >1mm from the resection margin, R1 as presence of tumor ≤1mm from the resection margin.
  * Number of harvested lymph nodes
  * Number of positive lymph nodes (infiltrated by tumor)
  * Tumor size, degree of differentiation, perineural and lymphovascular invasion
Differences in locoregional lymphadenectomy in patients with pancreatic adenocarcinoma | During surgery
  In a sub-cohort of patients with pancreatic adenocarcinoma, the number of harvested and positive lymph nodes (infiltrated by tumor) will be assessed and compared between the two groups.
Postoperative recurrence in patients with pancreatic adenocarcinoma | Postoperative Day 1 up to 5 years after surgery
  Patients with pancreatic adenocarcinoma who undergo resection in each arm will be followed postoperatively to document disease recurrence, defined as the re-presentation of measurable tumor after resection.
Postoperative survival in patients with pancreatic adenocarcinoma | Postoperative Day 1 up to 5 years after surgery
  Patients with pancreatic adenocarcinoma who undergo resection in each arm will be followed postoperatively to document overall survival, defined as the time between date of operation and date of death.
Perioperative costs | Postoperative Day 1 to Day 90
  Comparison of cost between the two groups, defined as the combination of intraoperative and postoperative costs, measured in US Dollars.

CONTACTS AND LOCATIONS:
Overall Officials: Baiyong Shen, PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nassour I, Winters SB, Hoehn R, Tohme S, Adam MA, Bartlett DL, Lee KK, Paniccia A, Zureikat AH. Long-term oncologic outcomes of robotic and open pancreatectomy in a national cohort of pancreatic adenocarcinoma. J Surg Oncol. 2020 Aug;122(2):234-242. doi: 10.1002/jso.25958. Epub 2020 Apr 29. PMID 32350882
- [Background] Shi Y, Jin J, Qiu W, Weng Y, Wang J, Zhao S, Huo Z, Qin K, Wang Y, Chen H, Deng X, Peng C, Shen B. Short-term Outcomes After Robot-Assisted vs Open Pancreaticoduodenectomy After the Learning Curve. JAMA Surg. 2020 May 1;155(5):389-394. doi: 10.1001/jamasurg.2020.0021. PMID 32129815
- [Background] Podda M, Gerardi C, Di Saverio S, Marino MV, Davies RJ, Pellino G, Pisanu A. Robotic-assisted versus open pancreaticoduodenectomy for patients with benign and malignant periampullary disease: a systematic review and meta-analysis of short-term outcomes. Surg Endosc. 2020 Jun;34(6):2390-2409. doi: 10.1007/s00464-020-07460-4. Epub 2020 Feb 18. PMID 32072286
- [Background] Zureikat AH, Beane JD, Zenati MS, Al Abbas AI, Boone BA, Moser AJ, Bartlett DL, Hogg ME, Zeh HJ 3rd. 500 Minimally Invasive Robotic Pancreatoduodenectomies: One Decade of Optimizing Performance. Ann Surg. 2021 May 1;273(5):966-972. doi: 10.1097/SLA.0000000000003550. PMID 31851003
- [Background] Girgis MD, Zenati MS, King JC, Hamad A, Zureikat AH, Zeh HJ, Hogg ME. Oncologic Outcomes After Robotic Pancreatic Resections Are Not Inferior to Open Surgery. Ann Surg. 2021 Sep 1;274(3):e262-e268. doi: 10.1097/SLA.0000000000003615. PMID 31663967
- [Background] Shi Y, Wang W, Qiu W, Zhao S, Wang J, Weng Y, Huo Z, Jin J, Wang Y, Deng X, Shen B, Peng C. Learning Curve From 450 Cases of Robot-Assisted Pancreaticoduocectomy in a High-Volume Pancreatic Center: Optimization of Operative Procedure and a Retrospective Study. Ann Surg. 2021 Dec 1;274(6):e1277-e1283. doi: 10.1097/SLA.0000000000003664. PMID 31651533
- [Background] Zhao W, Liu C, Li S, Geng D, Feng Y, Sun M. Safety and efficacy for robot-assisted versus open pancreaticoduodenectomy and distal pancreatectomy: A systematic review and meta-analysis. Surg Oncol. 2018 Sep;27(3):468-478. doi: 10.1016/j.suronc.2018.06.001. Epub 2018 Jun 4. PMID 30217304
- [Background] McMillan MT, Zureikat AH, Hogg ME, Kowalsky SJ, Zeh HJ, Sprys MH, Vollmer CM Jr. A Propensity Score-Matched Analysis of Robotic vs Open Pancreatoduodenectomy on Incidence of Pancreatic Fistula. JAMA Surg. 2017 Apr 1;152(4):327-335. doi: 10.1001/jamasurg.2016.4755. PMID 28030724
- [Background] Zureikat AH, Postlewait LM, Liu Y, Gillespie TW, Weber SM, Abbott DE, Ahmad SA, Maithel SK, Hogg ME, Zenati M, Cho CS, Salem A, Xia B, Steve J, Nguyen TK, Keshava HB, Chalikonda S, Walsh RM, Talamonti MS, Stocker SJ, Bentrem DJ, Lumpkin S, Kim HJ, Zeh HJ 3rd, Kooby DA. A Multi-institutional Comparison of Perioperative Outcomes of Robotic and Open Pancreaticoduodenectomy. Ann Surg. 2016 Oct;264(4):640-9. doi: 10.1097/SLA.0000000000001869. PMID 27433907
- [Derived] Jin J, Shi Y, Chen M, Qian J, Qin K, Wang Z, Chen W, Jin W, Lu F, Li Z, Wu Z, Jian L, Han B, Liang X, Sun C, Wu Z, Mou Y, Yin X, Huang H, Chen H, Gemenetzis G, Deng X, Peng C, Shen B. Robotic versus Open Pancreatoduodenectomy for Pancreatic and Periampullary Tumors (PORTAL): a study protocol for a multicenter phase III non-inferiority randomized controlled trial. Trials. 2021 Dec 27;22(1):954. doi: 10.1186/s13063-021-05939-6. PMID 34961558